CLINICAL TRIAL: NCT01022203
Title: Couples Treatment of PTSD in OEF/OIF Veterans
Brief Title: Comparison of Couple-Based PTSD Treatment and Couple-Based PTSD Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6756-R
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-10

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Couples Therapy; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Approach Therapy (Experimental): Couple-Based Intervention called Structured Approach Therapy provides skills training to couple so they can reduce PTSD.
  Interventions: Behavioral: Structured Approach Therapy
- PTSD Family Education (Active Comparator): Couple-Based Education called PTSD Family Education teaches couple about PTSD symptoms, related problems, and treatment.
  Interventions: Other: PTSD Family Education

INTERVENTIONS:
Behavioral: Structured Approach Therapy — The Structured Approach Therapy intervention includes education about the impact of PTSD on relationships; skills training to teach couples recognize and stop avoidance behavior; behavior activation training; emotion regulation training; and a couple-based intervention to teach Veterans with PTSD to identify and disclose trauma memories and related emotions to their partners. The couple is then trained to support disclosure while practicing empathic communication.
  Arms: Structured Approach Therapy
Other: PTSD Family Education — The PTSD Family Education intervention provides education for Veterans with PTSD and their partners explaining the signs and symptoms of PTSD; psychological problems that are comorbid with PTSD; and treatments for PTSD. Skills training and psychotherapy are not included.
  Arms: PTSD Family Education

SUMMARY:
The study is designed to evaluate the efficacy of a novel couple-based treatment for PTSD, called Structured Approach Therapy, to decrease PTSD and improve the marital and social functioning of Iraqi war Veterans and their partners. The effectiveness of couples therapy will be compared with the effectiveness of a couple-based educational intervention.

DETAILED DESCRIPTION:
The goal of the proposed study is to test the efficacy of a novel couple-based PTSD treatment, called Structured Approach Therapy, by randomly assigning 57 Iraqi war Veterans and their partners to either a 12-15 session Structured Approach Therapy program, or to a 12-15 session PTSD Family Education comparison condition. The efficacy of the two experimental conditions will be ascertained by obtaining measures of PTSD severity from Veterans and measures of relationship functioning and emotion regulation from Veterans and their partners prior to treatment, immediately after treatment, and three months after the last treatment session. The investigators will test the hypothesis that couples participating in Structured Approach Therapy will show significantly greater improvements on all three clinical outcome measures than couples participating in PTSD Family Education. These hypotheses will be tested with an intent-to-treat analysis using general linear mixed models with main effects of treatment, time (baseline, end of treatment, and 12 week follow-up), and treatment by time interactions to model the longitudinal trajectories of the outcome, separately for the Veterans and their partners. The objectives of the Structured Approach Therapy intervention are to decrease PTSD severity, improve relationship and family functioning, and decrease problems in emotion regulation in a group of young Veterans at risk for developing chronic PTSD, and to reduce emotional distress and relationship and family problems in their partners.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to at least one combat-related stressful event during combat deployment,
* Current diagnostic criteria for PTSD for that event, and
* Veteran is in a committed relationship and living with an opposite sex partner for at least six months.

Exclusion Criteria:

* Current psychotic symptoms in either partner,
* Current diagnosis of alcohol or drug dependence in either partner,
* History of recent physical assault/abuse,
* Currently receiving an evidence-based PTSD treatment (exposure-based or cognitive processing therapy)
* Currently receiving couples therapy or family therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic J Sautter, PhD, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sautter FJ, Glynn SM, Cretu JB, Senturk D, Vaught AS. Efficacy of structured approach therapy in reducing PTSD in returning veterans: A randomized clinical trial. Psychol Serv. 2015 Aug;12(3):199-212. doi: 10.1037/ser0000032. PMID 26213789
- [Result] Sautter FJ, Glynn SM, Becker-Cretu JJ, Senturk D, Armelie AP, Wielt DB. Structured Approach Therapy for Combat-Related PTSD in Returning U.S. Veterans: Complementary Mediation by Changes in Emotion Functioning. J Trauma Stress. 2016 Aug;29(4):384-7. doi: 10.1002/jts.22120. Epub 2016 Jul 29. PMID 27472747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-four subjects (12 couples) were lost or withdrew from the study after providing consent and participating in the pretreatment assessment, but before randomization to one of the two treatment conditions (Structured Approach Therapy or PTSD Family Education).
Groups:
- Structured Approach Therapy: Couple's Therapy Intervention
  Structured Approach Therapy: Couple's Therapy for PTSD
- PTSD Family Education: Educational Intervention.
  PTSD Family Education: Education about PTSD for couples.
Period: PreTreatment Assessment
Arm/Group | Structured Approach Therapy | PTSD Family Education
Started | 58 | 56
Completed | 58 | 56
Not Completed | 0 | 0
Period: Post Treatment Assessment
Arm/Group | Structured Approach Therapy | PTSD Family Education
Started | 58 | 56
Completed | 44 | 42
Not Completed | 14 | 14
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 0 | 2
Period: Follow-Up Assessment
Arm/Group | Structured Approach Therapy | PTSD Family Education
Started | 44 | 42
Completed | 42 | 40
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: These variables were entered into initial GLMM outcome models with no variable predicting outcome.
Groups:
- Arm 1: Couple's Therapy Intervention
  Structured Approach Therapy: Couple's Therapy for PTSD
- Arm 2: Educational Intervention.
  PTSD Family Education: Education about PTSD for couples.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Veterans Age | 33.71 (7.01) | 32.55 (6.16) | 33.12 (6.56)
  Partners Age | 32.25 (7.89) | 32.17 (7.68) | 32.21 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 56 | 56 | 112
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Psychological Functioning
Description: Clinician-Rated PTSD measured with the Clinician Administered PTSD Scale (Score range 0-133 with high scores indicating more severe PTSD); Self-Rated PTSD measured with the PTSD Checklist (Score range 17-85 with high scores indicating more severe PTSD).
Time Frame: Pre-Treatment, Post-treatment (12 weeks), Follow-up (12 weeks after post-treatment).
Population: Outcome data collected from 44 veterans who participated in Structured Approach Therapy and 42 Veterans who participated in PTSD Family Education.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Structured Approach Therapy: Veterans participate in pre-treatment assessment; post-treatment assessment within one week of the last study assessment, and a follow-up assessment 12 weeks after the last intervention session. Partners also participate but do not provide data.
- PTSD Family Education: Veterans participate in pre-treatment assessment; post-treatment assessment within one week week of the last study assessment, and a follow-up assessment 12 weeks after the last intervention session. Partners also participate but do not provide data.
Arm/Group | Structured Approach Therapy | PTSD Family Education
Number analyzed (Participants) | 44 | 42
units on a scale
  Vet Pre-treatment Clinician Administered PTSD Scal | 82.93 (3.31) | 82.93 (3.31)
  Vet Pre-treatment PTSD Checklist | 60.84 (2.12) | 60.81 (2.17)
  Vet Post-treatment Clinician Administered PTSD | 48.33 (3.71) | 72.59 (3.79)
  Vet Post-treatment PTSD Checklist | 42.16 (2.38) | 53.91 (2.48)
  Vet Followup Clinician Administered PTSD Scale | 44.64 (3.78) | 71.93 (3.86)
  Vet Followup PTSD Checklist | 39.54 (2.48) | 51.77 (2.53)
Statistical Analysis 1: Comparison: Structured Approach Therapy vs PTSD Family Education; Used Intent to Treat Analysis. General linear mixed models (GLMMs) with main effects of treatment (SAT and PFE), time (baseline, end of treatment, and 12 week follow-up), and treatment by time interactions to model the longitudinal trajectories of the outcomes, for veterans and their partners. Time was flexibly modeled. All available observations from each subject were utilized in the GLMM modeling; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Slope = .0001

2. Secondary Outcome: Relationship Functioning
Description: Relationship functioning is defined as relationship adjustment; measured with the Dyadic Adjustment Scale. The Dyadic Adjustment Scale scores range from 0-151 with high scores indicating high levels of relationship adjustment.
Time Frame: Pre-Treatment, Post-treatment (12 weeks), Follow-up (12 weeks after post-treatment).
Population: Data collected from 44 veterans participating in Structured Approach Therapy and 42 veterans participating in PTSD Family Education.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Structured Approach Therapy; PTSD Family Education: Pre-Treatment, Post-Treatment (12 weeks), Follow-up (12 weeks after post-treatment).
Arm/Group | Structured Approach Therapy | PTSD Family Education
Number analyzed (Participants) | 44 | 42
units on a scale
  Vet Pre-Trtmt Dyadic Adjustment Scale | 93.34 (3.53) | 101.82 (3.60)
  Vet Post-Trtmt Dyadic Adjustment Scale | 105.18 (3.84) | 101.77 (3.87)
  Vet Followup Dyadic Adjustment Scale | 106.76 (3.84) | 101.95 (3.91)
Statistical Analysis 1: Comparison: Structured Approach Therapy vs PTSD Family Education; Used Intent to Treat Analysis. General linear mixed models (GLMMs) with main effects of treatment (SAT and PFE), time (baseline, end of treatment, and 12 week follow-up), and treatment by time interactions to model the longitudinal trajectories of the outcomes for veterans. Time was flexibly modeled. All available observations from each subject were utilized in the GLMM modeling; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Slope = .004

3. Secondary Outcome: Emotion Regulation
Description: Measured with the Difficulties in Emotion Regulation Scale which measures severity of emotion regulation problems (Scores range from 36-125 with higher scores indicating higher levels of emotion regulation problems).
Time Frame: Pre-Treatment, Post-treatment (12 weeks), Follow-up (12 weeks after post-treatment).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Structured Approach Therapy | PTSD Family Education
Number analyzed (Participants) | 44 | 42
units on a scale
  Vet Pre-Trtmt Difficulties in Emotion Regulation | 106.6 (23.9) | 106.4 (22.4)
  Vet Post-Trtmt Difficulties in Emotion Regulation | 88.7 (24.4) | 106.4 (22.4)
  VetFollowup Difficulty in Emotion Regulation Scale | 87.29 (26.84) | 105.75 (25.99)
Statistical Analysis 1: Comparison: Structured Approach Therapy vs PTSD Family Education; General linear mixed models with main effects of treatment, time (baseline, end of treatment, and 12 week follow-up), and treatment by time interactions as described for previous analyses; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Structured Approach Therapy (SAT): Couple-Based Intervention called Structured Approach Therapy (SAT) provides skills training to couple so they can reduce PTSD.
  Structured Approach Therapy (SAT): Structured Approach Therapy (SAT) intervention includes education about the impact of PTSD on relationships; skills training to teach couples recognize and stop avoidance behavior; behavior activation training; emotion regulation training; and a couple-based intervention to teach veterans with PTSD to identify and disclose trauma memories and related emotions to their partners. The couple is then trained to support disclosure while practicing empathic communication.
- PTSD Family Education (PFE): Couple-Based Education called PTSD Family Education (PFE) teaches couple about PTSD symptoms, related problems, and treatment.
  PTSD Family Education (PFE): PTSD Family Education (PFE) provides education for veterans with PTSD and their partners explaining the signs and symptoms of PTSD; psychological problems that are comorbid with PTSD; and treatments for PTSD. Skills training and psychotherapy are not included.
Arm/Group | Structured Approach Therapy (SAT) | PTSD Family Education (PFE)
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 0/58 | 2/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Structured Approach Therapy (SAT) (N=58) | PTSD Family Education (PFE) (N=56)
Domestic violence (Psychiatric disorders) | 0 (0) | 2 (2) — Veteran and his spouse became intoxicated and veteran was violent with spouse. No serious injury and no medical treatment required. The spouse ended her relationship with the veteran.

LIMITATIONS AND CAVEATS:
The study's small sample size makes results preliminary and precludes formal hypothesis testing of mediating variables. Our report of decreased PTSD may reflect regression toward the mean.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes